CLINICAL TRIAL: NCT05298059
Title: The Effect of Photobiomodulation Therapy Associated With Casein Phosphopeptide-amorphous Calcium Phosphate Fluoride Paste on the Treatment of Post-home Whitening Tooth Sensitivity: a Randomized Clinical Trial
Brief Title: The Association of CPP-ACPF Associated With LASER in the Treatment of Tooth Sensitivity After at Home Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Clinical professor, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFPara05
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Sensitivity, Tooth
Keywords: Sensitivity, Tooth; Laser; Tooth Bleaching; Dentin Desensitizing Agents
MeSH Terms: conditions — Dentin Sensitivity | interventions — Clinical Trials Data Monitoring Committees

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind study, so that to blind study participants, all treatments were performed in exactly the same way. To simulate the CPP-ACPF paste, a paste without active ingredient was manipulated, but with the same color, texture and smell of the CPP-ACPF paste. To simulate the application of the laser, the operator performed the clinical procedure of applying the laser to three bridges of each tooth, but without activating it. The sound emitted by the laser at each point was simulated by a cell phone application.
  To blind the evaluator of the results, he only had access to the patient's name and sensitivity data, but he did not have access to the group to which the participant belonged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CPP-ACPF PASTE APLICATION (Placebo Comparator): Apply the cpp-acpf paste, at four different times (one each week of whitening treatment), for five minutes in each application and evaluate if it was able to reduce the sensitivity after home whitening with 22% carbamide peroxide.
  Interventions: Drug: CPP-ACPF
- Evaluate the effectiviness at home bleaching (No Intervention): To evaluate the effectiveness of at-home bleaching with 22% carbamide peroxide, with the help of the VITA Easyshade 4.0 spectrophotometer
- LASER APLICATION (Placebo Comparator): Apply the laser at four different times (one every week of whitening treatment), using the spectrum of infrared light with a wavelength of 808 nm with its active medium of Arsento Gallium and Aluminum (AsGaAl), at three points, one in the center of the crown of the tooth, another in the center of the cervical region and the last one in the incisal region, with the light beam directed apically, from all teeth to the second premolar of each upper and lower hemi-arch, with energy of of 1 Joule per point for 10 seconds. and evaluate if it was able to reduce the sensitivity after home whitening with 22% carbamide peroxide.
  Interventions: Radiation: Laser of low frequncy
- Associate the CPP-ACPF paste with the LASER (Placebo Comparator): Associate the CPP-ACPF paste with the LASER, following the same clinical protocol mentioned above and assess whether the association is more efficient than both treatments alone.
  Interventions: Radiation: Laser of low frequncy; Drug: CPP-ACPF

INTERVENTIONS:
Radiation: Laser of low frequncy — Apply the laser at three points on each tooth.
  Other Names: Therapy EC, DMC
  Arms: Associate the CPP-ACPF paste with the LASER; LASER APLICATION
Drug: CPP-ACPF — Apply MI paste plus for five minutes, in the vestibular surface os teeth. During this time patientes should be with closed mounth ad should not talk or to split.
  Other Names: MI paste plus
  Arms: Associate the CPP-ACPF paste with the LASER; CPP-ACPF PASTE APLICATION

SUMMARY:
Tooth whitening is a procedure that has been increasingly requested by patients around the world, whether at home or in office bleaching. Tooth sensitivity is the main side effect of bleaching. It have a great power to interfere negatively in the quality of life of those affected. According to the literature, about 51% of people who had at-home bleaching developed postoperative sensitivity.

The objective of this clinical, randomized, double-blind study is to evaluate the effectiveness of the association of casein phosphopeptides-fluoridated amorphous calcium phosphate with photobiomodulation in the treatment of tooth sensitivity after home bleaching, with 22% carbamide peroxide and also evaluate the effectiveness of at home bleaching through color analysis.

For develop this study, 50 patients will be selected, with no previous history of sensitivity, aged between 18 and 30 years. They will be divided into four treatment groups: PLACEBO group; CPP-ACPF group; LASER group; LASER+CPP-ACPF group.

Home bleaching treatment will use 22% carbamide peroxide. Patients should use two hours a day for 21 days. The desensitizing treatments will be applied in four moments, according to the group of each patient: before starting the bleaching treatment; after one week of the bleaching treatment; after two weeks of whitening treatment and after three weeks of whitening treatment.

Sensitivity will be assessed using a visual analogue scale (VAS), where patients should daily mark their pain level (from 0 to 10) on each side of the arcade. After the 21 days of treatment, they will receive a new VAS, to evaluate if was any sensitivity will occur during 30 days after the bleaching treatment.

In parallel with bleaching treatment and sensitivity treatment, the color analysis of teeth 13, 11, 21 and 23 will be performed, with the Vita Easyshade Advance 4.0 spectrophotometer, to monitor the bleaching performance, in each week. The first one will occur before starting the bleaching treatment (baseline) and a new measurement will be performed every week, together with the application of treatments for sensitivity.

The collected data will be tabulated in an Excel Microsoft Windows 2010) spreadsheet and analyzed in the Jamovi 1.6.23 (The Jamovi Project, 2020) software. For inter- and intra-group analysis of sensitivity values, the Repeated Measures statistical test will probably be used. For all statistical analyses, a significance level of 5% will be adopted.

DETAILED DESCRIPTION:
Tooth whitening is a procedure that has been increasingly requested by patients around the world, whether at home or in office bleaching. Tooth sensitivity is the main side effect of bleaching. It have a great power to interfere negatively in the quality of life of those affected. According to the literature, about 51% of people who had at-home bleaching developed postoperative sensitivity.

The objective of this clinical, randomized, double-blind study is to evaluate the effectiveness of the association of casein phosphopeptides-fluoridated amorphous calcium phosphate with photobiomodulation in the treatment of tooth sensitivity after home bleaching, with 22% carbamide peroxide and also evaluate the effectiveness of at home bleaching through color analysis.

Fifty patients will be selected, who will be divided into four treatment groups: PLACEBO group (will receive a LASER simulation and a manipulated paste without active ingredient to simulate the CPP-ACPF paste); CPP-ACPF group (will receive the CPP-ACPF folder and a LASER simulation); LASER group (will receive the LASER and a manipulated paste without active ingredient to simulate the CPP-ACPF paste); LASER+CPP-ACPF group (will receive the LASER and the CPP-ACPF folder). As it is a split-mouth study, each patient will receive two different types of treatment, one on each side of the arches, thus, the sample size of each group will be 25 patients (n=25).

The treatment with the CPP-ACPF paste (MI paste plus) will be carried out in the CPP-ACPF and LASER+CPP-ACPF groups, at the following times: before the bleaching treatment (T0), after one week of bleaching (T1), after two weeks of bleaching (T2), after three weeks of bleaching (T3). The application will be made on the buccal surfaces of the teeth, up to the second premolars, with the aid of a microbrush applicator (Microbrush, 3M Espe), for five minutes. Afterwards, patients will be instructed to spit out the excess and avoid ingesting anything for 30 minutes. In the PLACEBO group, this clinical protocol will be performed exactly, but using the paste without active ingredient.

The LASER and CPP-ACPF+FBM groups will receive the application of LASER (Therapy EC, DMC, São Carlos, SP, Brazil), using the infrared light spectrum with a wavelength of 808 nm with its active medium of Arsento Gallium and Aluminum (AsGaAl), at three points, one in the center of the crown of the tooth, another in the center of the cervical region and the last one in the incisal region, with the light beam directed apically, from all teeth to the second premolar of each hemi -upper and lower arch. The energy used was 1 Joule per point for 10 seconds.

While the PLACEBO and CPP-ACPF groups received a LASER simulation. The sounds emitted by the laser during its use will be simulated by a mobile application.

All study participants will receive a tube of bleaching agent (Whiteness Simple 22%, FGM, Joinville, Brazil) and will be instructed to apply a drop of the product on the vestibular surface of each tooth on the whitening tray (up to the second premolars) and use for two uninterrupted hours for 21 days.

Sensitivity will be assessed using a visual analogue scale (VAS), where patients should daily mark their pain level (from 0 to 10) on each side of the arcade. After the 21 days of treatment, they will receive a new VAS, to evaluate if was any sensitivity will occur during 30 days after the bleaching treatment.

In parallel with bleaching treatment and sensitivity treatment, the color analysis of teeth 13, 11, 21 and 23 will be performed, with the Vita Easyshade Advance 4.0 spectrophotometer, to monitor the bleaching performance, in each week. The first one will occur before starting the bleaching treatment (baseline) and a new measurement will be performed every week, together with the application of treatments for sensitivity.

The collected data will be tabulated in an Excel Microsoft Windows 2010) spreadsheet and analyzed in the Jamovi 1.6.23 (The Jamovi Project, 2020) software. For inter- and intra-group analysis of sensitivity values, the Repeated Measures statistical test will probably be used. For all statistical analyses, a significance level of 5% will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years;
* Good general and oral health;
* Sound incisors, canines and premolars;
* Prior whitening treatment;
* No hypersensitivity;

Exclusion Criteria:

* Patients undergoing fixed orthodontic treatment;
* Presence of periodontal disease;
* Presence of cracks or fractures;
* Presence of restorations and prostheses in anterior teeth;
* Extensive restorations in molars;
* Presence of gastroesophageal dysfunctions;
* Patients with severe internal dental darkening;
* Presence of exposed dentin.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Sensitivity assessment | Afeter 21 days of tooth whitening
  Aplly Repeated Measures ANOVA to analyze tooth sensitivity data reported by patients

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Federal University of Pará, Belém, Pará
  - Maria Eduarda Cardoso, Belém, Pará

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guanipa Ortiz MI, Alencar CM, Freitas De Paula BL, Alves EB, Nogueira Araujo JL, Silva CM. Effect of the casein phosphopeptide-amorphous calcium phosphate fluoride (CPP-ACPF) and photobiomodulation (PBM) on dental hypersensitivity: A randomized controlled clinical trial. PLoS One. 2019 Dec 2;14(12):e0225501. doi: 10.1371/journal.pone.0225501. eCollection 2019. PMID 31790452
- [Background] Dahl JE, Pallesen U. Tooth bleaching--a critical review of the biological aspects. Crit Rev Oral Biol Med. 2003;14(4):292-304. doi: 10.1177/154411130301400406. PMID 12907697
- [Background] Pontes M, Gomes J, Lemos C, Leao RS, Moraes S, Vasconcelos B, Pellizzer EP. Effect of Bleaching Gel Concentration on Tooth Color and Sensitivity: A Systematic Review and Meta-analysis. Oper Dent. 2020 May/Jun;45(3):265-275. doi: 10.2341/17-376-L. PMID 32396502
- [Background] de Vasconcelos AA, Cunha AG, Borges BC, Machado CT, dos Santos AJ. Tooth whitening with hydrogen/carbamide peroxides in association with a CPP-ACP paste at different proportions. Aust Dent J. 2012 Jun;57(2):213-9. doi: 10.1111/j.1834-7819.2012.01683.x. Epub 2012 Apr 4. PMID 22624764
- [Background] Huq NL, Myroforidis H, Cross KJ, Stanton DP, Veith PD, Ward BR, Reynolds EC. The Interactions of CPP-ACP with Saliva. Int J Mol Sci. 2016 Jun 9;17(6):915. doi: 10.3390/ijms17060915. PMID 27294918
- [Background] Szesz A, Parreiras S, Martini E, Reis A, Loguercio A. Effect of flowable composites on the clinical performance of non-carious cervical lesions: A systematic review and meta-analysis. J Dent. 2017 Oct;65:11-21. doi: 10.1016/j.jdent.2017.07.007. Epub 2017 Jul 17. PMID 28729119
- [Background] Chidchuangchai W, Vongsavan N, Matthews B. Sensory transduction mechanisms responsible for pain caused by cold stimulation of dentine in man. Arch Oral Biol. 2007 Feb;52(2):154-60. doi: 10.1016/j.archoralbio.2006.09.009. Epub 2006 Nov 15. PMID 17109813
- [Background] Splieth CH, Tachou A. Epidemiology of dentin hypersensitivity. Clin Oral Investig. 2013 Mar;17 Suppl 1(Suppl 1):S3-8. doi: 10.1007/s00784-012-0889-8. Epub 2012 Dec 7. PMID 23224064
- [Background] Pompeu DDS, de Paula BLF, Barros APO, Nunes SC, Carneiro AMP, Araujo JLN, Silva CM. Combination of strontium chloride and photobiomodulation in the control of tooth sensitivity post-bleaching: A split-mouth randomized clinical trial. PLoS One. 2021 Apr 28;16(4):e0250501. doi: 10.1371/journal.pone.0250501. eCollection 2021. PMID 33909659
- [Background] Sasaki RT, Arcanjo AJ, Florio FM, Basting RT. Micromorphology and microhardness of enamel after treatment with home-use bleaching agents containing 10% carbamide peroxide and 7.5% hydrogen peroxide. J Appl Oral Sci. 2009 Nov-Dec;17(6):611-6. doi: 10.1590/s1678-77572009000600014. PMID 20027436
- [Background] Hosseinpour S, Tuner J, Fekrazad R. Photobiomodulation in Oral Surgery: A Review. Photobiomodul Photomed Laser Surg. 2019 Dec;37(12):814-825. doi: 10.1089/photob.2019.4712. Epub 2019 Nov 21. PMID 31750798
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. PLoS Med. 2010 Mar 24;7(3):e1000251. doi: 10.1371/journal.pmed.1000251. PMID 20352064
- [Background] Gerritsen AE, Allen PF, Witter DJ, Bronkhorst EM, Creugers NH. Tooth loss and oral health-related quality of life: a systematic review and meta-analysis. Health Qual Life Outcomes. 2010 Nov 5;8:126. doi: 10.1186/1477-7525-8-126. PMID 21050499
- [Result] Sulieman M, Addy M, MacDonald E, Rees JS. The effect of hydrogen peroxide concentration on the outcome of tooth whitening: an in vitro study. J Dent. 2004 May;32(4):295-9. doi: 10.1016/j.jdent.2004.01.003. PMID 15053912
- [Result] Kielbassa AM, Maier M, Gieren AK, Eliav E. Tooth sensitivity during and after vital tooth bleaching: A systematic review on an unsolved problem. Quintessence Int. 2015 Nov-Dec;46(10):881-97. doi: 10.3290/j.qi.a34700. PMID 26396993
- [Result] Moosavi H, Arjmand N, Ahrari F, Zakeri M, Maleknejad F. Effect of low-level laser therapy on tooth sensitivity induced by in-office bleaching. Lasers Med Sci. 2016 May;31(4):713-9. doi: 10.1007/s10103-016-1913-z. Epub 2016 Mar 10. PMID 26964798
- [Result] Rezende M, Loguercio AD, Kossatz S, Reis A. Predictive factors on the efficacy and risk/intensity of tooth sensitivity of dental bleaching: A multi regression and logistic analysis. J Dent. 2016 Feb;45:1-6. doi: 10.1016/j.jdent.2015.11.003. Epub 2015 Dec 2. PMID 26612623
- [Result] Gojkov-Vukelic M, Hadzic S, Zukanovic A, Pasic E, Pavlic V. Application of Diode Laser in the Treatment of Dentine Hypersensitivity. Med Arch. 2016 Dec;70(6):466-469. doi: 10.5455/medarh.2016.70.466-469. PMID 28210023